CLINICAL TRIAL: NCT02929953
Title: Prevalence of Premature Birth History Among Type 1 Diabetes Mellitus (T1D) Patients and Characteristics of Premature Born Children Who Develop T1D Compared With Those Who do Not
Brief Title: Prematurity Prevalence Among T1D Patients and Its Characteristics Compared With Premature-born Non-diabetic Patients
Acronym: T1Dpremies
Status: Completed | Type: Observational
Sponsor: Assaf Harofeh MC (Other Government)
Collaborators: Shaare Zedek Medical Center (Other); Wolfson Medical Center (Other Government); Ziv Medical Center (Other); Schneider Children's Medical Center, Israel (Other); Tel-Aviv Sourasky Medical Center (Other Government); Maccabi Healthcare Services, Israel (Other); Kaplan Medical Center (Other); HaEmek Medical Center, Israel (Other); Soroka University Medical Center (Other); Rambam Health Care Campus (Other); Hadassah Medical Organization (Other)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Assaf-Harofeh Medical Center, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 183/13
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: premature birth; risk factor; type 1 diabetes mellitus; seasonality; prevalence; enteral feeding; immunomodulating medications; early onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes mellitus type 1: all T1DM patients in Israel, born during 2000-2013 and diagnosed prior to January 2015.
  chart review
  Interventions: Other: chart review
- Non-diabetic: non-diabetic general population born in Israel during 2000-2013, according to the Israeli Health Ministry's Birth Registry (IHMBR) chart review
  Interventions: Other: chart review

INTERVENTIONS:
Other: chart review — data from charts and from registries will be compared

SUMMARY:
The aims of this study are:

1. To assess the prevalence of prematurity, especially early prematurity, among T1D patients, and compare it to the prematurity prevalence among the non-diabetic general population in Israel.
2. To characterize epidemiological and clinical factors that differ between premature-born patients that developed T1D and those that have not, including the nutritional and therapeutic properties in NICU.

DETAILED DESCRIPTION:
A national cohort study, including linkage of data from 13 pediatric diabetes centers and Israeli National Registries, including all patients with T1D born during 1990-2013. Data collected includes: ethnicity, gestational age, birth season, age and season at T1DM diagnosis, and presence of autoimmunity in family. The prevalence of prematurity among T1D is compared to the non-diabetic general population registry of 2000-2013. Additional comparisons are between T1D patients born term and preterm, aimed to unveil specific influencing clinical and epidemiological factors.

In the latter part of the study, a multi-centered, paired case-control study is performed.

Preterm born T1D patients will be paired to matched non-diabetic children at a ratio of 3:1, according to medical center, sex, gestational week of birth, season and year of birth. Data collected includes: ethnicity, family history of autoimmune diseases, age and type of first enteral nutrition, and pharmacological exposures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with T1D
2. Patients treated in one of the 13 participating centers
3. For the case-control portion of the study, all children born between 1.1.1990-31.12.2013 and admitted to NICU medical centers that have been included in the original cohort portion
4. Patients for whom a complete medical record is available

Exclusion Criteria:

1. Lack of birth data
2. Unknown type of diabetes
3. For case control portion, an incomplete medical record/inadequate documentation

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All T1D patients in Israel, born during 1990-2013 and diagnosed prior to January 2015, time of data collection. Inclusion criteria included all patients diagnosed as T1D by a pediatric endocrinologist according to the American Diabetes Association criteria, and treated for their T1D with insulin. Patients are identified from registries of the 13 participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
prematurity prevalence among T1D patients | 1 years
  the number of premature born among those with type 1 diaetes compared to prematurity in health non diabetic population

SECONDARY OUTCOMES:
food exposure of premature who developed T1DM compared with prematures who did not develop diabetes | 1 years
  75 files of premies with T1DM will be ccompared to 225 charts of premies, non diabetic for age of food initiation
Medications exposure in premature who developed T1DM compared with prematures who did not develop diabetes | 1 years
  75 files of premies with T1DM will be ccompared to 225 charts of premies, non diabetic for age and type of drugs initiation

CONTACTS AND LOCATIONS:
Overall Officials: marianna Rachmiel, md, Principal Investigator — Assaf Haroffeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No
IPD data will not be available for anyone other than the PI and co-investigators.

REFERENCES:
- [Background] Blumenfeld O, Dichtiar R, Shohat T; Israel IDDM Registry Study Group (IIRSG). Trends in the incidence of type 1 diabetes among Jews and Arabs in Israel. Pediatr Diabetes. 2014 Sep;15(6):422-7. doi: 10.1111/pedi.12101. Epub 2013 Nov 27. PMID 24283719
- [Background] Egro FM. Why is type 1 diabetes increasing? J Mol Endocrinol. 2013 Jul 12;51(1):R1-13. doi: 10.1530/JME-13-0067. Print 2013. PMID 23733895
- [Background] De Curtis M, Rigo J. The nutrition of preterm infants. Early Hum Dev. 2012 Mar;88 Suppl 1:S5-7. doi: 10.1016/j.earlhumdev.2011.12.020. Epub 2012 Jan 17. PMID 22261289
- [Background] Working Group Of Pediatrics Chinese Society Of Parenteral And Enteral Nutrition, Working Group Of Neonatology Chinese Society Of Pediatrics, Working Group Of Neonatal Surgery Chinese Society Of Pediatric Surgery. CSPEN guidelines for nutrition support in neonates. Asia Pac J Clin Nutr. 2013;22(4):655-63. doi: 10.6133/apjcn.2013.22.4.21. PMID 24231027
- [Background] Kagohashi Y, Otani H. Role of nutritional factors at the early life stages in the pathogenesis and clinical course of type 1 diabetes. Biomed Res Int. 2015;2015:382165. doi: 10.1155/2015/382165. Epub 2015 Mar 26. PMID 25883958
- [Background] Ziegler AG, Pflueger M, Winkler C, Achenbach P, Akolkar B, Krischer JP, Bonifacio E. Accelerated progression from islet autoimmunity to diabetes is causing the escalating incidence of type 1 diabetes in young children. J Autoimmun. 2011 Aug;37(1):3-7. doi: 10.1016/j.jaut.2011.02.004. Epub 2011 Mar 3. PMID 21376535
- [Background] Jaberi-Douraki M, Liu SW, Pietropaolo M, Khadra A. Autoimmune responses in T1DM: quantitative methods to understand onset, progression, and prevention of disease. Pediatr Diabetes. 2014 May;15(3):162-74. doi: 10.1111/pedi.12148. PMID 24827702
- [Background] Walker WA. Initial intestinal colonization in the human infant and immune homeostasis. Ann Nutr Metab. 2013;63 Suppl 2:8-15. doi: 10.1159/000354907. Epub 2013 Nov 8. PMID 24217032
- [Background] Kemppainen KM, Ardissone AN, Davis-Richardson AG, Fagen JR, Gano KA, Leon-Novelo LG, Vehik K, Casella G, Simell O, Ziegler AG, Rewers MJ, Lernmark A, Hagopian W, She JX, Krischer JP, Akolkar B, Schatz DA, Atkinson MA, Triplett EW; TEDDY Study Group. Early childhood gut microbiomes show strong geographic differences among subjects at high risk for type 1 diabetes. Diabetes Care. 2015 Feb;38(2):329-32. doi: 10.2337/dc14-0850. Epub 2014 Dec 17. PMID 25519450
- [Background] Kostic AD, Gevers D, Siljander H, Vatanen T, Hyotylainen T, Hamalainen AM, Peet A, Tillmann V, Poho P, Mattila I, Lahdesmaki H, Franzosa EA, Vaarala O, de Goffau M, Harmsen H, Ilonen J, Virtanen SM, Clish CB, Oresic M, Huttenhower C, Knip M; DIABIMMUNE Study Group; Xavier RJ. The dynamics of the human infant gut microbiome in development and in progression toward type 1 diabetes. Cell Host Microbe. 2015 Feb 11;17(2):260-73. doi: 10.1016/j.chom.2015.01.001. Epub 2015 Feb 5. PMID 25662751
- [Background] Zeitlin J, Szamotulska K, Drewniak N, Mohangoo AD, Chalmers J, Sakkeus L, Irgens L, Gatt M, Gissler M, Blondel B; Euro-Peristat Preterm Study Group. Preterm birth time trends in Europe: a study of 19 countries. BJOG. 2013 Oct;120(11):1356-65. doi: 10.1111/1471-0528.12281. Epub 2013 May 24. PMID 23700966
- [Background] Soll RF, Edwards WH. Antibiotic use in neonatal intensive care. Pediatrics. 2015 May;135(5):928-9. doi: 10.1542/peds.2015-0707. No abstract available. PMID 25896842
- [Background] Li S, Zhang M, Tian H, Liu Z, Yin X, Xi B. Preterm birth and risk of type 1 and type 2 diabetes: systematic review and meta-analysis. Obes Rev. 2014 Oct;15(10):804-11. doi: 10.1111/obr.12214. Epub 2014 Jul 30. PMID 25073871
- [Background] Cardwell CR, Carson DJ, Patterson CC. Parental age at delivery, birth order, birth weight and gestational age are associated with the risk of childhood Type 1 diabetes: a UK regional retrospective cohort study. Diabet Med. 2005 Feb;22(2):200-6. doi: 10.1111/j.1464-5491.2005.01369.x. PMID 15660739
- [Background] Crump C, Winkleby MA, Sundquist K, Sundquist J. Risk of diabetes among young adults born preterm in Sweden. Diabetes Care. 2011 May;34(5):1109-13. doi: 10.2337/dc10-2108. Epub 2011 Mar 16. PMID 21411504
- [Background] Algert CS, McElduff A, Morris JM, Roberts CL. Perinatal risk factors for early onset of Type 1 diabetes in a 2000-2005 birth cohort. Diabet Med. 2009 Dec;26(12):1193-7. doi: 10.1111/j.1464-5491.2009.02878.x. PMID 20002469
- [Background] Capasso L, Borrelli A, Cerullo J, Pisanti R, Figliuolo C, Izzo F, Paccone M, Ferrara T, Lama S, Raimondi F. Role of immunoglobulins in neonatal sepsis. Transl Med UniSa. 2014 Dec 19;11:28-33. eCollection 2015 Jan-Apr. PMID 25674546
- [Background] Gritz EC, Bhandari V. The human neonatal gut microbiome: a brief review. Front Pediatr. 2015 Mar 5;3:17. doi: 10.3389/fped.2015.00017. eCollection 2015. PMID 25798435
- [Background] Arboleya S, Sanchez B, Milani C, Duranti S, Solis G, Fernandez N, de los Reyes-Gavilan CG, Ventura M, Margolles A, Gueimonde M. Intestinal microbiota development in preterm neonates and effect of perinatal antibiotics. J Pediatr. 2015 Mar;166(3):538-44. doi: 10.1016/j.jpeds.2014.09.041. Epub 2014 Oct 25. PMID 25444008
- [Background] Modi SR, Collins JJ, Relman DA. Antibiotics and the gut microbiota. J Clin Invest. 2014 Oct;124(10):4212-8. doi: 10.1172/JCI72333. Epub 2014 Oct 1. PMID 25271726
- [Background] Uusitalo U, Liu X, Yang J, Aronsson CA, Hummel S, Butterworth M, Lernmark A, Rewers M, Hagopian W, She JX, Simell O, Toppari J, Ziegler AG, Akolkar B, Krischer J, Norris JM, Virtanen SM; TEDDY Study Group. Association of Early Exposure of Probiotics and Islet Autoimmunity in the TEDDY Study. JAMA Pediatr. 2016 Jan;170(1):20-8. doi: 10.1001/jamapediatrics.2015.2757. PMID 26552054
- [Derived] Adar A, Shalitin S, Eyal O, Loewenthal N, Pinhas-Hamiel O, Levy M, Dally-Gottfried O, Landau Z, Zung A, Levy-Khademi F, Zangen D, Tenenbaum-Rakover Y, Rachmiel M. Prevalence of early and late prematurity is similar among pediatric type 1 diabetes patients and the general population. Diabetes Metab Res Rev. 2018 Jul;34(5):e2996. doi: 10.1002/dmrr.2996. Epub 2018 Mar 24. PMID 29471580